CLINICAL TRIAL: NCT00869895
Title: A Phase I Dose-Finding Study of E7050 Administered Orally to Patients With Advanced Solid Tumors
Brief Title: A Dose-Finding Study of E7050 Administered Orally to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7050-E044-101
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2012-11

CONDITIONS: Cancer
Keywords: Advanced solid tumors
MeSH Terms: conditions — Neoplasms | interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7050

INTERVENTIONS:
Drug: E7050 — Oral dosing starting at 100 mg once daily. After the MTD of once daily dosing has been determined, subsequent cohorts will be treated with a divided dosing schedule either twice or three times daily. The starting dose for this schedule will be an appropriate level below the MTD for once daily dosing.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of E7050 given orally in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years.
2. Histologically and/or cytologically confirmed metastatic solid tumors, that have progressed after treatment with approved therapies, or for which there are no standard effective therapies available.
3. Adequate bone marrow function.
4. Adequate renal function.
5. Adequate liver function.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Life expectancy > 3 months.
8. Be willing and able to comply with the study protocol, and can give written informed consent.

   Additional inclusion criterion for the additional 15 patients recruited to the expanded MTD cohort only:
9. At least one tumor lesion with diameter >= 2 cm measurable according to Modified RECIST.

Exclusion Criteria:

1. Any condition that may preclude oral intake or oral absorption, history of gastrointestinal malabsorption, or surgery involving gastro- and/or intestinal- anastomosis within 4 weeks prior to starting study drug.
2. Untreated or unstable known primary or metastatic central nervous system (CNS) tumors (stability shown by contrast-enhanced computed tomography or magnetic resonance imaging scans at least 8 weeks apart, with the most recent scan obtained within 28 days prior to starting study treatment).
3. Known human immunodeficiency virus (HIV), hepatitis B or C, or severe/uncontrolled infection or intercurrent illness (unrelated to tumor).
4. Prior surgery, radiotherapy, chemotherapy, biologic therapy or investigational drugs within 4 weeks prior to starting study drug. Prior immunotherapy, hormonal, or molecular targeted therapy within 2 weeks prior to starting study treatment (except gonadorelin analogue therapy for prostate cancer is allowed). (All acute toxicities related to prior treatments should have resolved).
5. Clinically significant cardiac impairment or unstable ischemic heart disease including a myocardial infarction within 6 months prior to starting study drug.
6. Requiring therapeutic anti-coagulant therapy (prophylactic dose of heparin or low molecular weight heparin is allowed).
7. Poorly controlled hypertension (defined as a change in hypertensive therapy within 3 months of starting study drug) or hypertension diagnosed at screening (defined as a repeat blood pressure measurement of 160/90 mmHg or higher).
8. Pregnancy or lactation. Female patients of childbearing potential must have a negative pregnancy test before inclusion into the study, and must agree to use medically acceptable methods of contraception (e.g. abstinence, or a double-barrier method [e.g. condom + spermicide, condom + diaphragm with spermicide], or IUD, or have a vasectomised partner) starting at Screening and throughout the entire study period and for 2 months after the last dose of study drug. Those female patients using hormonal contraceptives must also be using an additional approved method of contraception (as described previously) starting at Cycle 1 Day 1, and continuing throughout the entire study period and for 2 months after the last dose of study drug.

   Perimenopausal women must have been amenorrheic for at least 12 months; otherwise a pregnancy test is required.

   Male patients must agree to use contraceptive methods (e.g., abstinence, or a double-barrier method [e.g., condom + spermicide, condom + partner diaphragm with spermicide]).

   Additional exclusion criterion for the additional 15 patients recruited to the expanded MTD cohort only:
9. History of any malignancy other than the present malignancy (except treated non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose: the highest dose at which no more than 1 out of 6 patients experiences Dose Limiting Toxicity (DLT) during Cycle 1. | Weekly assessments during the first 4 weeks of treatment.

SECONDARY OUTCOMES:
DLTs and adverse events. | Weekly assessments during the first 4 weeks of treatment for DLTs and throughout the study for AEs.
Pharmacokinetics (blood and urine). | Weekly assessments of blood during Cycle 1 and every 2 weeks for subsequent cycles and of urine on Day 1 of Cycles 1 and 2.
Pharmacodynamics (blood). | Weekly assessments during Cycle 1, every 2 weeks on Cycle 2, and on Day 1 of subsequent cycles.
Best overall tumor response, duration of response and duration of stable disease assessed according to modified RECIST (Response Evaluation Criteria in Solid Tumors). | At Screening, between Days 21 and 28 of every even cycle, and at the Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Hanekom, Study Director — Eisai Limited
Locations (2):
- United Kingdom (2):
  - Christie Hospital, Manchester
  - Royal Marsden Hospital, Surrey